CLINICAL TRIAL: NCT01318096
Title: A Randomized, Pilot Estimation Study to Compare the Safety and Efficacy of Raltegravir+TDF+3TC Versus TDF+3TC+EFV in HBV/HIV Co-infected Patients
Brief Title: Safety and Efficacy of Raltegravir+TDF+3TC in HBV/HIV Co-infected Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yunnan AIDS Care Center (Other)
Responsible Party: Xi-cheng Wang, Yunnan Provincial Hospital of Infectious Diseases/Yunnan AIDS Care Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSD-38154
Record Dates: First submitted 2011-03-08; First posted 2011-03-18 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-03

CONDITIONS: HBV Coinfection; HIV Infections
Keywords: safety; efficacy; raltegravir; HBV/HIV co-infection
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Tenofovir; Lamivudine; efavirenz, lamivudine, tenofovir disoproxil fumarate drug combination; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A:Raltegravir + tenofovir+lamivudine (Experimental)
  Interventions: Drug: raltegravir and tenofovir and lamivudine
- B:Efavirenz+tenofovir+lamivudine (Active Comparator)
  Interventions: Drug: efavirenz+tenofovir+lamivudine

INTERVENTIONS:
Drug: raltegravir and tenofovir and lamivudine — raltegravir 400mg BID and tenofovir 300mg qd and lamivudine 300mg gd for 48 weeks
  Other Names: raltegravir: Isentress
  Arms: A:Raltegravir + tenofovir+lamivudine
Drug: efavirenz+tenofovir+lamivudine — efavirenz 600mg QN +tenofovir 300mg qd +lamivudine 300mg qd for 48 weeks
  Other Names: efavirenz: Sustiva
  Arms: B:Efavirenz+tenofovir+lamivudine

SUMMARY:
In this pilot study, the investigators would examine the safety and efficacy of integrase inhibitor-Raltegravir in the control of HIV/HBV co-infection.

DETAILED DESCRIPTION:
There are in total more than 72939 HIV infected people reported in Yunnan, the largest number for any province in China. About 800 HIV inpatients are admitted to our hospital every year, amongst them about 10% co-infected with HBV. HIV and HBV co-infection patients must receive two drugs active against both HIV and HBV, for example Tenofovir disoproxil fumarate (TDF)+ lamivudine (3TC) or TDF+FTC. TDF and 3TC are nucleotide analogues that can inhibit both HIV and HBV DNA polymerases (Dore, Cooper et al. 2004). Combination therapy could decrease drug resistance. In China, TDF is a second-line drug of the national free ART program; however FTC is not in the list of free drugs. There is likely higher risk of causing drug resistance in treating HBV or HIV infection with 3TC or TDF monotherapy than combination therapy.

Raltegravir inhibits the catalytic activity of HIV-1 integrase, and does not significantly inhibit human phosphoryl transferases including DNA polymerases α, β, and γ, and may have less adverse effects. In chronic HBV infection, HBV-DNA does integrate into human DNA which results in difficulty eradicating HBV from the patient's body.

In this pilot study, the investigators would examine the safety and efficacy of integrase inhibitor-Raltegravir in the control of HIV/HBV co-infection.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent
* HIV-1 infection, documented in patient medical record. Acceptable forms of documentation include positive HIV antibody or detectable HIV RNA
* HIV-1 antiretroviral therapy naïve
* Chronic HBV infection, defined as HBsAg positive >6 months. Both HBeAg positive and negative subjects will be eligible
* Detectable HBV DNA ( > 300 copies/ml)
* Serum alpha-fetoprotein (AFP) of ≤ 50 ng/ml within 4 weeks of study entry, or if elevated > 50 ng/ml, an imaging study demonstrating no evidence of hepatic tumor within 4 weeks of enrollment

Exclusion Criteria:

* Allergy or sensitivity to study drug
* Pregnancy, breastfeeding or unwillingness/inability to adhere to contraceptive methods for the duration of the study (Female study volunteers must not participate in a conception process (e.g., active attempt to become pregnant). If participating in sexual activity that could lead to pregnancy, the female study volunteer must use the following forms of contraception while receiving study-specific medication(s) and for 30 days after stopping the medication. One of the following methods MUST be used appropriately: (1)Condoms* (male or female) with or without a spermicidal agent; (2)Diaphragm or cervical cap with spermicide; (3)IUD; (4)Hormonal-based method.Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV transmission.
* Prisoners or subjects who are incarcerated
* Receipt of the following drugs with anti-HBV activity within 90 days prior to study entry or anticipated receipt during the course of the study including: ADV, telbivudine, alpha interferon, and other investigational agents with anti-HBV activity
* Active opportunistic infection
* Other causes of chronic liver disease identified (autoimmune hepatitis, haemochromatosis, Wilsons disease, alfa-1-antitrypsin deficiency)
* Concurrent malignancy requiring cytotoxic chemotherapy
* Decompensated or Child's C cirrhosis
* Any other condition which in the opinion of the investigator might interfere with compliance or outcome of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-07 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | In 48 weeks (from baseline to study completion at 48 weeks)
  The investigators will collect the adverse events at every follow-up, and record them in CRFs. All AEs during the study will be analyzed according to the type, frequency and severity.

SECONDARY OUTCOMES:
Change of plasma HIV-1 RNA levels | week 0,24 and 48
Change of Peripheral blood CD4 cell counts | week 0,4,8,12,24,36 and 48
Change of plasma HBV-DNA levels | week 0,12,24,36,and 48
Change of serum total bilirubin levels（TBI） | week 0,2,4,8,12,24,36 and 48
Proportion of subjects with HBeAg seroconversion (HBeAg loss and presence of anti HBe) | week 0,12,24,36,and week 48
Emergence of drug resistance mutations, if appropriate | week 0, 24 and 48
Paired liver biopsy comparison according to inflammatory activity and fibrosis score | week 0 and 48
Change of serum alanine aminotransferase levels (ALT) | week 0,2,4,8,12,24,36 and 48
Change of serum aspartate aminotransferase levels (AST) | week 0,2,4,8,12,24,36 and 48
Change of blood urine nitrogen levels (BUN) | week 0,2,4,8,12,24,36 and 48
Change of serum creatinine levels (SCr) | week 0,2,4,8,12,24,36 and 48
Change of blood haemoglobin levels (HB) | week 0,2,4,8,12,24,36 and 48
Change of white blood cell counts (WBC) | week 0,2,4,8,12,24,36 and 48
Change of blood platelet counts (PLT) | week 0,2,4,8,12,24,36 and 48
Change of urine protein levels | week 0,2,4,8,12,24,36 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Xi Wang, M.D., Principal Investigator — Yunnan Provincial Hospital of Infectious Diseases/Yunnan AIDS Care Center
Locations (1):
- Yunnan Provincial Hospital of Infectious Diseases/Yunnan AIDS Care Center, Kunming, Yunnan Provice, China